CLINICAL TRIAL: NCT03367546
Title: Haploidentical Donor T-cell Replete Allogeneic Hematopoietic Cell Transplant Following Reducing Intensity Conditioning for Patients With Selected High Risk Non-Malignant Disease
Brief Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation (HaploHCT) Following Reduced Intensity Conditioning (RIC) for Selected High Risk Non-Malignant Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study no longer needed
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS101; MT2017-30 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease; Thalassemia; High Risk Hematologic Disorders; Cerebral Adrenoleukodystrophy; Inherited Metabolic Disorders
Keywords: SCD; cALD
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rATG, FLU/CY/TBI, & Thiotepa (Experimental): Anti-Thymocyte Globulin - Rabbit (rATG), Fludarabine (Fludara), Cyclophosphamide (Cytoxan, Neosar), Total Body Irradiation (TBI), & Thiotepa
  Interventions: Procedure: Blood and Marrow Transplant

INTERVENTIONS:
Procedure: Blood and Marrow Transplant — Reduced intensity conditioning (RIC) with rabbit ATG, fludarabine, cyclophosphamide, thiotepa and low dose (2 Gy) total body irradiation followed by T-cell replete, unmanipulated, haploidentical related donor stem cell transplant (HaploHCT) and post-transplant cyclophosphamide (PTCy)

SUMMARY:
This is a Phase II study for the use of T-cell replete reduced intensity conditioning (RIC) haploidentical donor allogeneic hematopoietic cell transplantation (HaploHCT) for individuals with high-risk non-malignant diseases who lack a suitable HLA-matched sibling donor.

ELIGIBILITY:
Inclusion Criteria:

* Sickle Cell Disease (SCD)

  * If diagnosis of SCD must meet one or more of the following disease characteristics:
  * Stroke, CNS hemorrhage or a neurologic event lasting longer than 24 hours, or abnormal cerebral MRI or cerebral arteriogram or MRI angiographic study and impaired neuropsychological testing
  * Acute chest syndrome with a history of recurrent hospitalizations or exchange transfusions
  * Recurrent vaso-occlusive pain 3 or more episodes per year for 3 years or more years or recurrent priapism,
  * Impaired neuropsychological function and abnormal cerebral MRI scan
  * Stage I or II sickle lung disease,
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate [GFR] 30-50% of the predicted normal value)
  * Bilateral proliferative retinopathy and major visual impairment in at least one eye
  * Osteonecrosis of multiple joints with documented destructive changes
  * Requirement for chronic transfusions
  * RBC alloimmunization
* Transfusion Dependent Alpha- or Beta-Thalassemia
* Other Non-Malignant Hematologic Disorders:

Transfusion dependent or involve other potential life-threatening cytopenias, including but not limited to Paroxysmal Nocturnal Hemoglobinuria, Glanzmann's Thrombasthenia, Severe Congenital Neutropenia and Shwachman-Diamond Syndrome

* cALD

  * Diagnosis of ALD by abnormal plasma very long chain fatty acid (VLCFA) profile or ABCD1 gene mutation
  * Cerebral disease on MRI
  * Absence of a Major Functional Disability (cortical blindness, loss of communication, wheelchair dependence) on the ALD Neurologic Function Scale
* Other inherited metabolic disorders:

Any other inherited metabolic disorder for which alloHCT is indicated and for whom, in the opinion of the treating physician, the patient's best treatment option is with a haploidentical donor following non-myeloablatve conditioning.

* Age, Performance Status, Consent

  * Age: 0-55 years
  * Performance Status: Karnofsky ≥ 70%, Lansky play score ≥ 70
  * Consent: voluntary written consent (adult or parental/guardian)
* Adequate Organ Function

  * Renal: Creatinine <2.0 mg/dl for adults or glomerular filtration rate > 50 ml/min for children
  * Hepatic: Bilirubin and ALT <3 times the upper limit of institutional normal
  * Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction > 40%.

Exclusion Criteria:

* Availability of a suitable HLA-matched related donor
* Uncontrolled infection
* Pregnant or breastfeeding
* HIV positive

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Neutrophil Recovery | Day 42
  Incidence of neutrophil recovery by day +42

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
  Incidence of overall survival at 1 year
Primary Graft Failure (neutropenic and non-neutropenic) | Day 42
  Incidence of primary graft failure (neutropenic and non-neutropenic) by day +42

CONTACTS AND LOCATIONS:
Overall Officials: Christen L Ebens, MD, MPH, Principal Investigator — University of Minnesota - Pediatrics Blood and Marrow Transplant
Locations (1):
- Masonic Caner Center at University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03367546/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03367546/ICF_001.pdf